CLINICAL TRIAL: NCT02744443
Title: Leucine Supplementation in Young Subjects Undergoing Resistance Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: LeucineUSP
Record Dates: First submitted 2016-04-12; First posted 2016-04-20 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Leucine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Leucine (Experimental): Leucine supplementation (10 g/d)
  Interventions: Dietary Supplement: Leucine
- Placebo (Placebo Comparator): Placebo supplementation (alanine, 10 g/d)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Leucine
  Arms: Leucine
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Leucine supplementation could be useful to support muscle anabolism. This study aims to investigate the effects of leucine supplementation on muscle mass and muscle strength in young subjects undergoing resistance training.

ELIGIBILITY:
Inclusion Criteria:

* training experience > 12 months
* no previous use of anabolic steroids
* no diagnosed diseases or injuries at the time of recruitment
* one-maximum repetition strength (1-RM) in leg press ≥ 3.5 and ≤ 5.0 times the body weight

Exclusion Criteria:

* use of creatine or beta-alanine supplements for the last 3 months
* use of protein or aminoacids supplements for the last 1 month
* engagement in specific dietary restrictions
* engagement in competitive sports

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
muscle cross-sectional area | 12 weeks
  B-mode ultrasound

SECONDARY OUTCOMES:
muscle strength | 12 weeks
  One repetition maximum (1RM) on 45º leg press machine and Muscular Endurance Test on 45º leg press machine

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No